CLINICAL TRIAL: NCT02301325
Title: Project 1, Study 2: The Combined Impact of Nicotine Replacement and Spectrum Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: U54 DA031659-P1S2; 1U54DA031659-01 (NIH)
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.03 mg Nicotine Cigarette (Other): Participants will be assigned to smoke 0.03 mg nicotine Spectrum cigarettes
  Interventions: Behavioral: Smoking research cigarettes with or without NRT
- 0.03 mg Nicotine Cigarette and NRT (Other): Participants will be assigned to smoke 0.03 mg nicotine Spectrum cigarettes and use nicotine replacement patches.
  Interventions: Behavioral: Smoking research cigarettes with or without NRT
- 0.80 mg Nicotine Cigarette (Other): Participants will be assigned to smoke 0.80 mg nicotine Spectrum cigarettes.
  Interventions: Behavioral: Smoking research cigarettes with or without NRT
- 0.80 mg Nicotine Cigarette and NRT (Other): Participants will be assigned to smoke 0.80 mg nicotine Spectrum cigarettes and use nicotine replacement patches.
  Interventions: Behavioral: Smoking research cigarettes with or without NRT

INTERVENTIONS:
Behavioral: Smoking research cigarettes with or without NRT

SUMMARY:
Project 1, Study 2 will evaluate the impact of very low nicotine content cigarettes with and without transdermal nicotine on cigarettes smoked per day, nicotine exposure, discomfort/dysfunction, other health-related behaviors, nicotine/tobacco dependence, biomarkers of tobacco exposure, intention to quit, compensatory smoking, other tobacco use, cigarette characteristics, cue reactivity, cardiovascular function, perceived risk and cue reactivity. The investigators will also consider differences between conditions in compliance with product use and the ability to abstain from smoking when provided a financial incentive for abstinence.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. Smoke an average of at least five cigarettes per day for the last year with no periods of continuous abstinence longer than 30 days.
3. Breath CO levels > or = 10 ppm (if < 10 ppm, then NicAlert Strip = 6)
4. Fulfills need for participants in the required strata (menthol status)

Exclusion Criteria:

1. Intention to quit smoking in the next 30 days
2. Currently seeking treatment for smoking cessation
3. Currently using nicotine replacement therapies or other pharmacotherapies as cessation aid (intermittent use acceptable)
4. Significant prior adverse reaction to nicotine replacement as determined by the licensed medical professional.
5. A quit attempt in the past 30 days resulting in greater than 3 days of abstinence
6. Using other tobacco products more than 9 days in the past 30 days
7. Significant unstable medical conditions (any significant change in a serious medical condition occurring during the past 3 months including cardiovascular disease, COPD, and cancer, as determined by the licensed medical professional)
8. Significant unstable psychiatric conditions (any significant change in psychiatric symptoms during the past 3 months as determined by the licensed medical professional)
9. Schizophrenia and schizoaffective disorder
10. Positive toxicology screen for any of the following drugs: marijuana, cocaine, opiates, methadone, benzodiazepines, barbiturates, amphetamines, methamphetamines, and PCP

    * Participants with valid prescriptions for any toxicology results will not be excluded.
11. Breath alcohol level > 0.01
12. Binge drinking alcohol (more than 9 days in the past 30 days, 4/5 drinks in a 2 hour period (female/male))
13. Pregnant, trying to become pregnant or breastfeeding
14. Smoking 'roll your own cigarettes' exclusively
15. Currently taking any one of the following medications:

    * Phenytoin [Brand Name: Dilantin]
    * Carbamazepine [Brand Name: Tegretol, Carbatrol, Equetro, Epitol]
    * Oxcarbazepine [Brand Name: Trileptal]
    * Primidone [Brand Name: Mysoline]
    * Phenobarbital
    * Bendamustine [Brand Name: Treanda]
    * Clopidogrel [Brand Name: Plavix]
    * Clozapine [Brand Name: Clozaril, FazaClo]
    * Erlotinib [Brand Name: Tarceva]
    * Flecainide [Brand Name: Tambocor]
    * Fluvoxamine [Brand Name: Luvox]
    * Irinotecan [Brand Name: Camptosar]
    * Olanzapine [Brand Name: Zyprexa]
    * Ropinirole [Brand Name: Requip]
    * Tacrine [Brand Name: Cognex]
    * Theophylline [Brand Name: Theo Dur]
    * Estradiol
16. CO reading >80 ppm
17. Systolic BP greater than or equal to 160

    * Participants failing for blood pressure will be allowed to re-screen once.
18. Diastolic BP greater than or equal to 100

    * Participants failing for blood pressure will be allowed to re-screen once.
19. Systolic BP below 90

    * Participants failing for blood pressure will be allowed to re-screen once.
20. Diastolic BP below 50

    * Participants failing for blood pressure will be allowed to re-screen once.
21. Heart rate greater than or equal to 105 bpm

    * Participants failing for heart rate will be allowed to re-screen once.
22. Heart rate lower than 45 bpm

    * Participants failing for heart rate will be allowed to re-screen once.
23. Indicating any suicidal ideation in the past month or suicide attempts in the past 5 years (if within the past 6-10 years, LMP approval required).
24. Inability to independently read and comprehend the consent form and other written study materials and measures.
25. Having participated in a research study during the past three months in which the participant:

    * Smoked a cigarette that was not his/her usual brand cigarette for more than one day
    * Used any tobacco products beyond normal use for more than one day
    * Used any nicotine replacement products or smoking cessation medications for more than one day
26. Having participated in Project 1, Study 1 (PRO11060292)
27. Having participated in Project 1, Study 1C (PRO14040384)
28. Household member enrolled in the study concurrently
29. Significant prior adverse reactions to adhesives or latex
30. Participant has a condition that interferes/does not allow for the collection of eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Cigarettes Smoked Per Day | Six Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Donny, Ph.D., Principal Investigator — Professor, University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Smith TT, Koopmeiners JS, Tessier KM, Davis EM, Conklin CA, Denlinger-Apte RL, Lane T, Murphy SE, Tidey JW, Hatsukami DK, Donny EC. Randomized Trial of Low-Nicotine Cigarettes and Transdermal Nicotine. Am J Prev Med. 2019 Oct;57(4):515-524. doi: 10.1016/j.amepre.2019.05.010. PMID 31542129